CLINICAL TRIAL: NCT06607809
Title: Association of Inflammatory Markers (ICC, MCVL) With Anti PD-1 Antibody Nivolumab Response: Evaluating Biomarkers for Predicting Immunotherapy Success in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Inflammatory Markers (ICC, MCVL) and Nivolumab Response: Predicting Immunotherapy Success in Metastatic RCC
Acronym: IMNR
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Heves Sürmeli, Consultant, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: 2024/010.99/6/9
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: RCC; Nivolumab; inflammatory marker; ICC; MCVL
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study is an observational study aimed at investigating the potential of new inflammatory markers to predict treatment response in patients with metastatic renal cell carcinoma (mRCC) undergoing anti-PD-1 antibody nivolumab therapy. Specifically, the study focuses on evaluating how well the Cumulative Inflammatory Index (ICC) and Mean Corpuscular Volume/Lymphocyte Ratio (MCVL) can predict the response to nivolumab treatment and the progression of the disease.

The participant group consists of patients aged 18 and older who have been diagnosed with metastatic renal cell carcinoma. Inflammatory markers were monitored at regular intervals throughout the treatment period.

The primary endpoints of the study are as follows:

1. Progression-Free Survival (PFS): To determine how long nivolumab treatment can halt disease progression.
2. Overall Survival (OS): To assess the overall survival of participants following treatment.
3. Disease Control Rate (DCR): To evaluate the disease control rates (stable disease, partial response, complete response) at 3, 6, and 12 months of Nivolumab treatment.

This study aims to deeply analyze the impact of inflammatory markers such as ICC and MCVL on disease progression and treatment response, determining to what extent these markers serve as predictors of treatment success. Additionally, it explores how these markers can be utilized in personalized treatment strategies to improve therapeutic outcomes.

DETAILED DESCRIPTION:
This observational study investigates the potential of new inflammatory markers to predict treatment response in patients with metastatic renal cell carcinoma (mRCC) undergoing anti-PD-1 antibody nivolumab therapy. The study specifically aims to evaluate how well the Cumulative Inflammatory Index (ICC) and Mean Corpuscular Volume/Lymphocyte Ratio (MCVL) can predict the response to nivolumab treatment and the progression of the disease.

Detailed Characteristics of the Participants:

Age Range: The participants cover a wide age range, from young adults to elderly individuals.

Gender and General Health Status: The gender of the participants is not specified, but all participants are adults diagnosed with metastatic renal cell carcinoma. Most have previously undergone treatment for renal cancer, and their disease has metastasized.

Histological Subtypes: The majority of participants have clear cell renal cell carcinoma (clear cell RCC). Other histological subtypes, including papillary, chromophobe, and sarcomatoid types, are also represented.

Metastasis Status: A significant proportion of the participants show metastasis to multiple organs. These metastases are most commonly found in the lungs, bones, brain, and liver.

Blood Parameters: Throughout the treatment, the blood values of the participants were regularly monitored. These parameters include white blood cells (WBC), red blood cells (RBC), hemoglobin (HGB), hematocrit (HCT), mean corpuscular volume (MCV), platelets (PLT), neutrophils, and lymphocytes.

Inflammatory Markers: The study tracks inflammatory markers such as the Cumulative Inflammatory Index (ICC) and Mean Corpuscular Volume/Lymphocyte Ratio (MCVL) in participants. These markers are believed to play an important role in the progression of the disease and the response to treatment.

Primary Endpoints of the Study:

Progression-Free Survival (PFS): The ability of nivolumab treatment to halt the progression of the disease over time is assessed.

Overall Survival (OS): The overall survival of participants following treatment is analyzed.

Disease Control Rate (DCR): The disease control rates (stable disease, partial response, complete response) at various time points during nivolumab treatment are evaluated.

Study Objective:

The primary aim of this study is to analyze the impact of inflammatory markers such as ICC and MCVL on disease progression and treatment response. Additionally, it seeks to explore how these markers can predict treatment success and be used in personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

Age: Participants must be ≥18 and ≤87 years old. Diagnosis: Patients must have been diagnosed with metastatic renal cell carcinoma (mRCC).

Treatment: Only patients receiving nivolumab treatment for metastatic renal cell carcinoma are included.

Consent: Written informed consent was obtained from all participants

Exclusion Criteria:

Other Active Cancers: Patients with concurrent active malignancies were excluded from the study.

Prior Immunotherapy Treatment: Patients who had previously received any form of immunotherapy (anti-PD-1, anti-PD-L1, or similar immunological agents) were excluded.

Uncontrolled Systemic Diseases: Patients with severe, uncontrolled systemic diseases (e.g., significant cardiovascular, pulmonary, or liver diseases) were not included in the study.

Active Infections: Patients with serious active infections, such as active tuberculosis, HIV infection, or chronic hepatitis B or C, were excluded.

Pregnancy and Breastfeeding: Pregnant or breastfeeding women were not eligible for inclusion in the study.

Immunodeficiency or Immunosuppressive Therapy: Patients with immunodeficiency or those receiving immunosuppressive therapy (e.g., corticosteroids) were excluded from the study.

Ages: 19 Years to 87 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients aged 18 and older diagnosed with metastatic renal cell carcinoma (mRCC). All participants are receiving nivolumab, an anti-PD-1 antibody, as part of their treatment for metastatic disease. Most patients have clear cell carcinoma, though other subtypes like papillary and sarcomatoid carcinoma are included.Patients have metastases in organs such as the lungs, bones, brain, and liver. The study monitors inflammatory markers, including the Cumulative Inflammatory Index (ICC) and Mean Corpuscular Volume/Lymphocyte Ratio (MCVL), at key time points. These biomarkers are evaluated for their role in predicting treatment response and disease progression, focusing on progression-free survival and overall survival in this population.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 3rd Month
  Progression-free survival (PFS) was assessed to determine if the disease had progressed, using disease control rates as a reference.
Progression-Free Survival | 6th Month
  Progression-free survival (PFS) was assessed to determine if the disease had progressed, using disease control rates as a reference.
Progression-Free Survival | 12th Month
  Progression-free survival (PFS) was assessed to determine if the disease had progressed, using disease control rates as a reference.
Disease Control Rate (DCR) | 3rd month
  The disease control rate (DCR) was evaluated to assess the response to treatment, including the rates of stable disease, partial response, and complete response.
Disease Control Rate (DCR) | 6th month
  The disease control rate (DCR) was evaluated to assess the response to treatment, including the rates of stable disease, partial response, and complete response.
Disease Control Rate (DCR) | 12th month
  The disease control rate (DCR) was evaluated to assess the response to treatment, including the rates of stable disease, partial response, and complete response.
Overall Survival | 3rd month
  Overall Survival (OS) was assessed to evaluate the survival status of the patients following treatment initiation.
Overall Survival | 6th month
  Overall Survival (OS) was assessed to evaluate the survival status of the patients following treatment initiation.
Overall Survival | 12th month
  Overall Survival (OS) was assessed to evaluate the survival status of the patients following treatment initiation.

SECONDARY OUTCOMES:
Changes in Inflammatory Markers (ICC) | 3rd month
  Inflammatory markers (ICC) will be regularly monitored, and any changes in these markers during treatment will be evaluated.
Changes in Inflammatory Markers (ICC) | 6th month
  Inflammatory markers (ICC) will be regularly monitored, and any changes in these markers during treatment will be evaluated.
Changes in Inflammatory Markers (ICC) | 12th month
  Inflammatory markers (ICC) will be regularly monitored, and any changes in these markers during treatment will be evaluated.
Changes in Inflammatory Markers (MCVL) | 3rd month
  Inflammatory markers (MCVL) will be regularly monitored, and any changes in these markers during treatment will be evaluated.
Changes in Inflammatory Markers (MCVL) | 6th month
  Inflammatory markers (MCVL) will be regularly monitored, and any changes in these markers during treatment will be evaluated.
Changes in Inflammatory Markers (MCVL) | 12th month
  Inflammatory markers (MCVL) will be regularly monitored, and any changes in these markers during treatment will be evaluated.
Immune-related adverse events (irAEs) | 3rd month
  Immune-related adverse events (irAEs) will be tracked, and the frequency and severity of these side effects will be assessed.
Immune-related adverse events (irAEs) | 6th month
  Immune-related adverse events (irAEs) will be tracked, and the frequency and severity of these side effects will be assessed.
Immune-related adverse events (irAEs) | 12th month
  Immune-related adverse events (irAEs) will be tracked, and the frequency and severity of these side effects will be assessed.
Response Based on Metastatic Sites | 3rd month
  The response to treatment in different metastatic sites (lungs, bones, brain, etc.) will be evaluated.
Response Based on Metastatic Sites | 6th month
  The response to treatment in different metastatic sites (lungs, bones, brain, etc.) will be evaluated.
Response Based on Metastatic Sites | 12th month
  The response to treatment in different metastatic sites (lungs, bones, brain, etc.) will be evaluated.
Evaluation of Neutrophil-Lymphocyte Ratio | 3rd month
  other blood parameters ( Neutrophil-Lymphocyte Ratio) will be analyzed for their potential to predict treatment success.
Evaluation of Neutrophil-Lymphocyte Ratio | 6th month
  other blood parameters ( Neutrophil-Lymphocyte Ratio) will be analyzed for their potential to predict treatment success.
Evaluation of Neutrophil-Lymphocyte Ratio | 12th month
  other blood parameters (Neutrophil-Lymphocyte Ratio) will be analyzed for their potential to predict treatment success.
Evaluation of Platelet-Lymphocyte Ratio | 3rd month
  other blood parameters (Platelet-Lymphocyte Ratio) will be analyzed for their potential to predict treatment success.
Evaluation of Platelet-Lymphocyte Ratio | 6th month
  other blood parameters (Platelet-Lymphocyte Ratio) will be analyzed for their potential to predict treatment success.
Evaluation of Platelet-Lymphocyte Ratio | 12th month
  other blood parameters (Platelet-Lymphocyte Ratio) will be analyzed for their potential to predict treatment success.

CONTACTS AND LOCATIONS:
Overall Officials: Heves Surmeli, MD, Principal Investigator — Health University Kartal Dr. Lütfi Kirdar City Hospital
Locations (1):
- Health Science University Kartal Dr. Lütfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)